CLINICAL TRIAL: NCT04584749
Title: Lidocaine as an Anesthetic Adjuvant in Upper Abdominal Laparoscopic Surgery
Brief Title: Lidocaine as an Anesthetic Adjuvant in Liver and Gastric Laparoscopic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Guillem Pla Escriva, Anesthetist, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROTOCOL LIDO
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: a phase IV, randomized, double-blind, two-arm, parallel-group clinical research trial
Who Masked: Participant, Investigator
Masking Description: Patients will be randomized in a 1: 1 ratio to one of two treatment groups: Lidocaine or Placebo.
  To preserve the masking of the study, the list with the recruited patients will be sent weekly to an independent researcher from IDIBGI, who will be in charge of providing the names and numbers of the medical records to the pharmacy service.
  The randomization process has been carried out using the PASS 16.0.4 program. Only the Pharmacy staff will know the randomization tables and codes. The main investigator will have the emergency codes in case of need
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIDOCAINE (Experimental): 2% lidocaine will be administered as a bolus during anesthetic induction equivalent to 1.5 mg / kg of lidocaine. After induction, an intravenous infusion will be started at 0.1 ml / kg / h of the study preparation, equivalent to 2mg / kg / h of lidocaine.
  The study medication will be prepared in a 20 ml syringe for induction and two 50 ml syringes for anesthetic maintenance containing 2% Lidocaine as assigned by the patient. The syringes prepared by the pharmacy will be identical in all cases, with a label specifying the title of this test and the identification number of the patient
  Interventions: Drug: Lidocaine Iv
- PLACEBO (Placebo Comparator): 0.9% physiological saline will be used as placebo, and it will be administered as a bolus during anesthetic induction . After induction, an intravenous infusion will be started at 0.1 ml / kg / h of the study preparation, equivalent to 2mg / kg / h of lidocaine/placebo.
  The study medication will be prepared in a 20 ml syringe for induction and two 50 ml syringes for anesthetic maintenance containing Physiological Serum as assigned by the patient. The syringes prepared by the pharmacy will be identical in all cases, with a label specifying the title of this test and the identification number of the patient
  Interventions: Drug: Lidocaine Iv

INTERVENTIONS:
Drug: Lidocaine Iv — 2% lidocaine or 0.9% physiological saline will be used as placebo, and it will be administered as a bolus during anesthetic induction equivalent to 1.5 mg / kg of lidocaine. After induction, an intravenous infusion will be started at 0.1 ml / kg / h of the study preparation, equivalent to 2mg / kg / h of lidocaine.
  20 ml syringe for induction and two 50 ml syringes for anesthetic maintenance containing 2% Lidocaine .

SUMMARY:
The aim is to analyze the effect of intravenous lidocaine administration on postoperative opioid use in patients undergoing upper abdominal cancer surgery. Specifically, those patients undergoing gastric cancer surgery and liver cancer surgery using a laparoscopic approach

DETAILED DESCRIPTION:
In a recent Cochrane Library review, despite the apparent positive results reported by intravenous administration of lidocaine as a perioperative analgesic adjuvant, the quality of the evidence is low, since the studies carried out to date present small samples, great variability in the designs and different surgical techniques studied.

More studies will be needed to help improve the grade and quality of evidence in the management of acute postoperative pain and its role in opioid sparing, an especially beneficial effect in tumor pathology For this reason, the investigators have designed a randomized, double-blind, phase IV clinical trial with two treatment arms, parallel groups, in which 96 patients who underwent liver and gastric cancer surgery through laparoscopic approach participated.

This study will include 2 different population groups: patients undergoing liver cancer surgery and patients undergoing gastric cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age scheduled for gastric or liver cancer surgery through a laparoscopic approach at the University of Girona Dr Josep Trueta.
* Accept and sign the informed consent

Exclusion Criteria:

* decline participating in the study at any stage of its development.
* History of allergic or adverse reactions to Amide-type anesthetics.
* Pregnancy or lactation period
* Diagnosis of Child-Pugh stage B or C liver failure.
* Acute renal failure (GFR <60 ml / min).
* Concomitant treatment with opioids for chronic pain.
* Any condition that, in the clinical judgment of the researchers, may interfere with the object of the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 Hours
  o evaluate the effect of intravenous lidocaine on postoperative pain after laparoscopic upper abdominal cancer surgery, analyzing postoperative opioid consumption

SECONDARY OUTCOMES:
Incidence of nausea and vomiting | 24 hours
  Analyze the incidence of nausea and vomiting, paralytic ileus, time of return to oral diet and hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Pla, MD, Principal Investigator — Hospital Dr Josep Trueta
Locations (1):
- Hospital Dr Josep Trueta, Girona, Spain

IPD SHARING:
Plan to Share IPD: No